CLINICAL TRIAL: NCT00958542
Title: Prospective Study of Scoliosis in Children With Cerebral Palsy
Brief Title: Prospective Study of Cerebral Palsy Scoliosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is coordinated by the Harms Study Group. It is already registered on this website
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H08-00897
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Cerebral Palsy; Scoliosis
Keywords: cerebral palsy; scoliosis; children
MeSH Terms: conditions — Cerebral Palsy; Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical Arm (Experimental): Surgical intervention for correction of scoliotic or kyphotic curvatures of the spine will include either the posterior approach or the anterior + posterior approach, with either the unit or custom rod, depending on the choice of the surgeon.
  Interventions: Procedure: Surgical fusion
- Non-Surgical Arm (No Intervention): Non-Surgical No intervention - Includes patients who have either refused to have surgery or have not been recommended to have surgery at this point. These patients will continue to be monitored closely, however, will not receive any other intervention.

INTERVENTIONS:
Procedure: Surgical fusion — Surgical intervention for correction of scoliotic or kyphotic curvatures of the spine will include either the posterior approach or the anterior + posterior approach, with either the unit or custom rod, depending on the choice of the surgeon.
  Arms: Surgical Arm

SUMMARY:
This is a prospective, multi-centre study that will be looking at two groups of males and females over the course of their operative treatment for cerebral palsy (CP) scoliosis and the years following that treatment. The first group the study will be looking at is those individuals who undergo surgery for CP Scoliosis. The second group will be those individuals who do not undergo surgical treatment for CP Scoliosis, either because the family declines surgery or surgery is not recommended during the course of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8 and 18 years
* Diagnosis of Cerebral Palsy with total body involvement
* Coronal curve greater than 40 degrees OR a kyphotic curve greater than 50 degrees on sitting film will be included
* Growing rod treatment will also be included

Exclusion Criteria:

* Previous operated scoliotic spine deformity
* Diagnosis of Rett's Syndrome
* Concomitant lower extremity surgery (within 3 months of spinal fusion)
* Cornelia de Lange Syndrome or any pervasive genetic disorder whose effects are due to much more than the static cortical injury
* Ambulatory spastic diplegic without upper extremity impairment or speech, swallowing or other involvement

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of pre- and post- operative x-rays | 1 year

SECONDARY OUTCOMES:
Gross motor function, physical data, past medical history, seizure status, pain and medications, sitting ability, activity level, clinical photos, quality of life questionnaires, data regarding surgery and hospital stay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Firoz Miyanji, Dr., Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada